CLINICAL TRIAL: NCT06019364
Title: Transfusion av Helblod - Egenskaper Hos Produkten Och Effekt av Transfusion Hos Patienter
Brief Title: Transfusion of Whole Blood in Acute Bleeding
Acronym: HEPEP
Status: Enrolling by invitation | Type: Observational
Sponsor: Sofia Ramström (Other)
Responsible Party: Sponsor-Investigator, Sofia Ramström, Associated Professor, Örebro University, Sweden
Organization: Örebro University, Sweden (Other)
Other Study IDs: 280695
Record Dates: First submitted 2023-07-12; First posted 2023-08-31 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Blood Transfusion; Acute Bleeding
MeSH Terms: interventions — Exchange Transfusion, Whole Blood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples without DNA retained from the patient (plasma and serum)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Whole blood transfusion — Transfusion of whole blood in a situation with acute bleeding according to routine practice.

SUMMARY:
Blood collected from blood donors is routinely divided into its different components, red blood cells, plasma and platelets. These components are stored under different storage conditions and their maximum storage time before transfusion is different. Platelets are stored at a maximum of 7 days and at a temperature of 22°C to best preserve their function.

Research has been conduction on blood stored and transfused as whole blood (without separation into the various components), particularly in situations of acute trauma. Region Örebro län will therefore start transfusion of whole blood in such situations. The whole blood units will be stored at 4°C for a maximum of 14 days. This means that the platelets will be stored at a lower temperature than standard and for a longer time period. The research on how this will affect platelet function is limited.

This project aims to determine how the patients are affected regarding coagulation, hemolysis, renal function, immunisation, transfusion reactions and the effect of substances released from the blood cells in the whole blood units during the storage period and if there is an impact on mortality.

DETAILED DESCRIPTION:
Blood collected from blood donors is routinely divided into its different components, red blood cells, plasma and platelets. These components are stored under different storage conditions and their maximum storage time before transfusion is different. Platelets are stored at a maximum of 7 days and at a temperature of 22°C to best preserve their function.

Platelets function is to contribute to the formation of a clot to stop and prevent bleeding. Previous studies has shown that this might be affected if they are stored refrigerated. Exactly how they are affected is not known and when this occurs during the storage period.

Research has been conduction on blood stored and transfused as whole blood (without separation into the various components), particularly in situations of acute trauma. Region Örebro län will therefore start transfusion of whole blood in such situations. The whole blood units will be stored at 4°C for a maximum of 14 days. This means that the platelets will be stored at a lower temperature than standard and for a longer time period. The research on how this will affect platelet function is limited.

Since transfusion of refrigerated whole blood is a new procedure this project aims to determine how the patients are affected regarding coagulation, hemolysis, renal function, immunisation, transfusion reactions and the effect of substances released from the blood cells in the whole blood units during the storage period and if there is an impact on mortality.

Patients requiring transfusion with a whole blood due to an acute situation with bleeding will be enrolled. Blood samples will be taken from the patients for analysis directly before the transfusion and at various time points after the transfusion. Clinical variables of importance to interpret the effect of the whole blood transfusion will be registered as well as basic information such as sex, age, height, weight, blood group and type of injury causing the bleeding, treatment etc.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute bleeding
* Transfused with whole blood at the time of the acute bleeding episode

Exclusion Criteria:

* Patients where vital information lacking needed to interpret data (i.e. blood cell count)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with acute bleeding that are transfused with whole blood at the time of the acute bleeding episode.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 day mortality
  Death within 30 days following the transfusion of whole blood
Effect of the whole blood transfusion on coagulation | All transfusions occuring within 24 hours post transfusion of the whole blood unit
  Requirement for other transfusions
Bleeding | All transfusions occuring within 24 hours post transfusion of the whole blood unit
  Bleeding following transfusion of the whole blood unit

SECONDARY OUTCOMES:
Hemolysis | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 2, Day 5, Day 30
  Hemolysis at various time points in conjunction to the whole blood transfusion
Platelet count | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 2, Day 5, Day 30
  Platelet count at various time points in conjunction to the whole blood transfusion
Red blood cell count | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 2, Day 5, Day 30
  Red blood cell count at various time points in conjunction to the whole blood transfusion
APTT, a marker of coagulation capacity | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of APTT at various time points in conjunction to the whole blood transfusion
PT, a marker of coagulation capacity | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of PT at various time points in conjunction to the whole blood transfusion
Anti-thrombin, a marker of coagulation capacity | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of anti-thrombin at various time points in conjunction to the whole blood transfusion
Fibrinogen, a marker of of coagulation capacity | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of fibrinogen at various time points in conjunction to the whole blood transfusion
Electrolytes | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Electrolytes at various time points in conjunction to the whole blood transfusion
Creatinine, a marker of of renal function | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of Creatinine at various time points in conjunction to the whole blood transfusion
GFR, a marker of renal function | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of GFR at various time points in conjunction to the whole blood transfusion
Urea, a measure of renal function | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of urea at various time points in conjunction to the whole blood transfusion
sP-selectin, a soluble marker of platelet activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of sP-selectin at various time points in conjunction to the whole blood transfusion
PF4, a soluble marker of platelet activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of PF4 at various time points in conjunction to the whole blood transfusion
MMP9, a soluble marker of platelet activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of MMP9 at various time points in conjunction to the whole blood transfusion
sCD40L, a soluble marker of platelet activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of sCD40L at various time points in conjunction to the whole blood transfusion
sGPV, a soluble marker of platelet activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of sGPV at various time points in conjunction to the whole blood transfusion
sGPVI, a soluble marker of platelet activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of sGPVI at various time points in conjunction to the whole blood transfusion
SCUBE1, a soluble marker of platelet activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of SCUBE1 at various time points in conjunction to the whole blood transfusion
TSP1, a soluble marker of platelet activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of TSP1 at various time points in conjunction to the whole blood transfusion
CRP, a marker of inflammation activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of CRP at various time points in conjunction to the whole blood transfusion
Serum amyloid A (SAA), a marker of inflammation activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of Serum amyloid A at various time points in conjunction to the whole blood transfusion
sTNFR1, a marker of inflammation activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of sTNFR1 at various time points in conjunction to the whole blood transfusion
sTNFR2, a marker of inflammation activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of sTNFR2 at various time points in conjunction to the whole blood transfusion
D-dimer, a marker of coagulation activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of D-dimer at various time points in conjunction to the whole blood transfusion
vWF, a marker of coagulation activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of vWF at various time points in conjunction to the whole blood transfusion
TAT, a marker of coagulation activation | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of TAT at various time points in conjunction to the whole blood transfusion
RANTES, a bio modulating substance | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of RANTES at various time points in conjunction to the whole blood transfusion
VEGF, a bio modulating substance | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of VEGF at various time points in conjunction to the whole blood transfusion
IFN-gamma, a bio modulating substance | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of IFN-gamma at various time points in conjunction to the whole blood transfusion
TNF-alfa, a bio modulating substance | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of TNF-alfa at various time points in conjunction to the whole blood transfusion
IL-7, a bio modulating substance | Day 0-pre transfusion, Day 0-post transfusion, Day 1, Day 5 and Day 30
  Analysis of IL-7 at various time points in conjunction to the whole blood transfusion
Immunisation | Within 30 days post transfusion
  Occurence of immunisation following transfusion of the whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Ramström, Ass. Prof, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No